CLINICAL TRIAL: NCT02703441
Title: FoodnGo - Empower: A Feasibility Study
Brief Title: FoodnGo-Empower: A Feasibility Study of Physical Activities and Nutrition of Older Patients by the Use of Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Tachista (Unknown)
Responsible Party: Principal Investigator, Tove Lindhardt Damsgaard, senior researcher, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-O-FNG-2015-1
Record Dates: First submitted 2015-03-17; First posted 2016-03-09 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Malnutrition; Physical Activity
MeSH Terms: conditions — Malnutrition; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention: Tablet computer (Experimental): Patients from the local municipality, planned to be discharged to a rehabilitation stay at the municipality training centre receive a tablet computer. The patient will be introduced to the tablet and informed about the nutritional and mobilisation intervention based on his/her individual needs and preferences. The patient and the research assistant will jointly prepare an individual plan for nutrition and physical activity The patient uses the tablet for ordering meals, registering dietary intake, viewing his/her instruction videos for the activity programme and registering physical activity during hospital admission and at the training centre up to 6 weeks after discharge from hospital.
  Interventions: Other: Tablet computer
- Control group (No Intervention): Patients in the control group receive usual care during their hospital stay and after discharge at the municipality training centre. Data are recorded at baseline and 6 and 12 weeks after discharge.

INTERVENTIONS:
Other: Tablet computer — Patients randomized to the intervention group will receive a tablet computer with an app-like software solution supporting nutrition and physical activity. The patients operate the computer and order their meals from the hospital menu; register dietary intake, and receive feedback informing about their current status for protein and energy intake. Likewise, the patients use small series of brief videos instructing in daily life activities for strengthening their muscles. After this, they register their performed activities and will receive informing and motivating feedback. Nudging and prompting is part of the solution.
  Other Names: Malnutrition and physical activity
  Arms: Intervention: Tablet computer

SUMMARY:
The research and innovation programme Food´n´Go - Empower aims to develop, test and implement health technology solutions for active involvement and increased empowerment of elderly patients and their relatives solving well-known problem areas as malnutrition and inactivity.

The prototype was developed in 2013. The project is a collaboration between departement of internal medicine in Copenhagen University Hospital, one local municipality and a private it-company. The technology is a tablet computer, used by elderly patients to order and register food intake during hospitalization. The tablet is also used to get inspiration for physical activities during hospital admission and after discharge and for registration of physical activities.

The aim of this study is to test if an adjusted version of the Food´n´Go technology through active involvement of the elderly patient can prevent weightloss and loss of muscle strength during hospitalization and after discharge.

DETAILED DESCRIPTION:
Welfare and health technology are often directed at solving problems and meeting the needs of societies' most vulnerable groups often not familiar with computers.

The research and innovation programme Food´n´Go - Empower aims to develop, test and implement health technology solutions for involvement and increased empowerment of elderly patients and their relatives. The focus is on frequent issues for this group of patients, in this phase focusing on nutrition and physical activity. Later, the solution will include pain management, management of sleep problems, medication management, prevention of confusion and coordination of the treatment and care course across sectorial borders. The technology is a tablet- computer, operated by the patient by means of a number of app-like software applications.

In the summer 2013 the programme received a grant from the Capitol Region's Public-Private-Innovation (OPI) pool for design and development of the prototype. In 2014 the prototype for nutrition was tested in a feasibility study. Usability and acceptability was tested in the patients' own home, as well as the effect of the nutrition intervention, after discharge from hospital (see protocol 10/16/2014).

The results were promising, and the aim is now to test the technology for supporting both nutrition and physical activity across sectorial boundaries. The elderly patient will operate the tablet during admission and after discharge, continuing the efforts aimed at nutrition and physical activity during the stay at a rehabilitation centre 5 to 6 weeks after discharge. The working hypothesis is: Functional ability and nutritional status will be stabilized or improved, and readmissions and dependency of municipal services will be reduced.

The aim of this study is:

1. to test if an adjusted version of the Food´n´Go technology through active involvement of the elderly patient can prevent weight loss and loss of muscle strength during hospitalization and after discharge
2. to develop and test the technology in relation to stability, applicability and acceptability

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years old admitted to Department of Internal Medicine
* Planned to be discharged to a temporary stay at the municipality training centre
* Body Mass Index ≤ 20
* Patient experienced problems with solving daily physical activities
* Minimal Mental State Examination (MMSE) ≥24
* Able to operate the computer
* Able to collaborate in the physical activities
* Has a relative who is willing to be supportive

Exclusion Criteria:

* Terminal patients
* Patients who are not able to communicate or do not understand danish

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in lean body-mass | Baseline, 6 weeks and 12 weeks
  DEXA scanning,

SECONDARY OUTCOMES:
Change in muscle strength | baseline, 6 and 12 weeks
  handgrip strength
Change in muscle strength | baseline, 6 and 12 weeks
  chair-stand-test
Change in weight | baseline, 6 and 12 weeks
Change in BMI | baseline, 6 and 12 weeks
Change in Health related Quality of Life | baseline, 6 and 12 weeks
  EQ5D (European Quality 5Dimensions Scale)
Change in signs of depression | Baseline, 6 and 12 weeks
  Geriatric Depression Scale 5 (GDS5)
Number of days to first readmission | 24 weeks
  Danish National Patient Register
Mortality | 24 weeks
  Danish National Patient Register

OTHER OUTCOMES:
Physical activity | 12 weeks
  Registered by the patient at the computer
Dietary intake | 12 weeks
  Registered by the patient at the computer
Technology functionality | 12 weeks
  Research assistant observes and registers problems
Technology stability | 12 weeks
  Research assistant observes and registers problems
Technology acceptability | 12 weeks
  Qualitative interviews with patients and relatives

CONTACTS AND LOCATIONS:
Overall Officials: Tove L. Damsgaaard, Ph.D., Principal Investigator — Herlev Hospital
Locations (1):
- Department of Internal Medicine, Copenhagen University Herlev, Herlev, Denmark